CLINICAL TRIAL: NCT00696020
Title: Randomised, Double-Blind, Parallel Group Study to Assess the Efficacy and Safety of 4 Weeks of Once Daily Treatment of 3 Doses of Orally Inhaled BI 1744 CL, Each in Fixed Dose Combination With 5 Microgram Tiotropium Bromide (Delivered by the Respimat Inhaler) Compared With 5 Microgram Tiotropium Bromide Monoproduct (Delivered by the Respimat Inhaler) in Patients With COPD
Brief Title: Combination of Orally Inhaled BI1744CL/Tiotropium Bromide in Patients With Chronic Obstructive Pulmonary Disease ( COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237.4; EudraCT No: 2007-005087-26
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- BI 1744 CL low dose/tiotropium bromide (Experimental): BI 1744 CL low dose plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: BI 1744 CL/tiotropium bromide fixed dose combination; Device: Respimat® Inhaler
- BI1744CL medium dose/tiotropium bromide (Experimental): BI 1744 CL medium dose plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: BI 1744 CL/tiotropium bromide fixed dose combination; Device: Respimat® Inhaler
- BI 1744 CL high dose/tiotropium bromide (Experimental): BI 1744 CL high dose plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: BI 1744 CL/tiotropium bromide fixed dose combination; Device: Respimat® Inhaler
- tiotropium bromide (Experimental): tiotropium bromide; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Interventions: Drug: tiotropium bromide; Device: Respimat® Inhaler

INTERVENTIONS:
Drug: BI 1744 CL/tiotropium bromide fixed dose combination — BI 1744 CL plus tiotropium bromide fixed dose combination; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Arms: BI 1744 CL high dose/tiotropium bromide; BI 1744 CL low dose/tiotropium bromide; BI1744CL medium dose/tiotropium bromide
Drug: tiotropium bromide — tiotropium bromide; Solution for inhalation via Respimat® Inhaler (A5); Oral inhalation
  Arms: tiotropium bromide
Device: Respimat® Inhaler

SUMMARY:
The primary objective of this study is to determine the optimum dose(s) of BI 1744 CL administered with 5 micrograms tiotropium bromide solution for inhalation, delivered by the Respimat inhaler, once daily for four weeks in patients with chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

1. All patients must sign an informed consent consistent with ICH-GCP guidelines prior to participation in the trial, which includes medication washout and restrictions
2. All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

   Patients must have relatively stable airway obstruction with a post-bronchodilator FEV1 greater or equal 30% of predicted normal and <80% of predicted normal and a post-bronchodilator FEV1 / FVC <70% at Visit 1
3. Male or female patients, 40 years of age or older
4. Patients must be current or ex-smokers with a smoking history of more than 10 pack years
5. Patients must be able to perform technically acceptable pulmonary function tests and PEF measurements, and must be able to maintain records (Patient Daily e-Diary) during the study period as required in the protocol
6. Patients must be able to inhale medication in a competent manner from the Respimat inhaler and from a metered dose inhaler (MDI).

Further inclusion criteria apply

Exclusion Criteria:

1. Patients with a significant disease other than COPD
2. Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis;
3. Patients with a history of asthma or a total blood eosinophil count >= 600/mm3.
4. Patients with any of the following conditions:a diagnosis of thyrotoxicosis, a diagnosis of paroxysmal tachycardia (>100 beats per minute), a marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTcF* interval > 450 ms), a history of additional risk factors for Torsade de Pointes (TdP) (e.g. heart failure, hypokalemia, family history of Long QT Syndrome)
5. Patients with any of the following conditions:a history of myocardial infarction within 1 year of screening visit (Visit 1), a diagnosis of clinically relevant cardiac arrhythmia, known active tuberculosis, a malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years, a history of life-threatening pulmonary obstruction, a history of cystic fibrosis, clinically evident bronchiectasis, a history of significant alcohol or drug abuse
6. Patients who have undergone thoracotomy with pulmonary resection
7. Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
8. Pregnant or nursing women
9. Women of childbearing potential not using two effective method of birth control (one barrier and one non-barrier). Female patients will be considered to be of childbearing potential unless surgically sterilised by hysterectomy or bilateral tubal ligation, or post-menopausal for at least two years
10. Patients who have previously been randomized in this study or are currently participating in another study
11. Patients who are unable to comply with pulmonary medication restrictions prior to randomization
12. Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening Visit

Further exclusion criteria apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (37):
- United States (22):
  - 1237.4.0118 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1237.4.0103 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1237.4.0115 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1237.4.0105 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1237.4.0110 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1237.4.0117 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1237.4.0104 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1237.4.0120 Boehringer Ingelheim Investigational Site, Edina, Minnesota
  - 1237.4.0112 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1237.4.0119 Boehringer Ingelheim Investigational Site, Saint Charles, Missouri
  - 1237.4.0114 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1237.4.0102 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1237.4.0111 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1237.4.0106 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.4.0107 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1237.4.0123 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 1237.4.0122 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1237.4.0109 Boehringer Ingelheim Investigational Site, New Braunfels, Texas
  - 1237.4.0108 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1237.4.0116 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1237.4.0121 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1237.4.0101 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Canada (8):
  - 1237.4.0203 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1237.4.0201 Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - 1237.4.0202 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.4.0205 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.4.0208 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1237.4.0206 Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
  - 1237.4.0204 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 1237.4.0207 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Germany (7):
  - 1237.4.4903 Boehringer Ingelheim Investigational Site, Berlin
  - 1237.4.4907 Boehringer Ingelheim Investigational Site, Erfurt
  - 1237.4.4902 Boehringer Ingelheim Investigational Site, Gauting
  - 1237.4.4908 Boehringer Ingelheim Investigational Site, Halle
  - 1237.4.4906 Boehringer Ingelheim Investigational Site, Neuruppin
  - 1237.4.4904 Boehringer Ingelheim Investigational Site, Rüdersdorf
  - 1237.4.4901 Boehringer Ingelheim Investigational Site, Weinheim

REFERENCES:
- [Derived] Maltais F, Hamilton A, Voss F, Maleki-Yazdi MR. Dose Determination for a Fixed-Dose Drug Combination: A Phase II Randomized Controlled Trial for Tiotropium/Olodaterol Versus Tiotropium in Patients with COPD. Adv Ther. 2019 Apr;36(4):962-968. doi: 10.1007/s12325-019-00911-y. Epub 2019 Mar 6. PMID 30843141

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A randomised, double-blind, parallel group study. Each patient received their randomised treatment for 28 days.
Groups:
- 5 µg Tiotropium: Oral inhalation of Tiotropium fixed dose 5 µg (2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium+Olodaterol 5/2 μg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 2 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 1.0 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium+Olodaterol 5/5 μg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium+Olodaterol 5/10 μg: Oral inhalation of fixed dose combination (FDC) of Tiotropium 5 µg and Olodaterol 10 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
Period: Overall Study
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Started | 90 | 89 | 93 | 88
Completed | 86 | 87 | 90 | 84
Not Completed | 4 | 2 | 3 | 4
Not completed — Adverse Event | 3 | 1 | 2 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Other not stated above | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS). The TS included all randomized patients who received at least 1 dose of study medication.
Groups:
- Tiotropium+Olodaterol 5/2 μg: Oral inhalation of FDC of Tiotropium 5 µg and Olodaterol 2 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 1.0 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium+Olodaterol 5/5 μg: Oral inhalation of FDC of Tiotropium 5 µg and Olodaterol 5 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 2.5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Tiotropium+Olodaterol 5/10 μg: Oral inhalation of FDC of Tiotropium 5 µg and Olodaterol 10 µg (Tiotropium: 2.5 µg per actuation and Olodaterol: 5 µg per actuation), 2 puffs from the Respimat inhaler, once daily, in the morning.
- Total: Total of all reporting groups
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg | Total
Number analyzed (Participants) | 90 | 89 | 93 | 88 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.87 (8.50) | 64.44 (9.18) | 64.19 (9.59) | 62.66 (8.86) | 63.30 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 33 | 45 | 39 | 164
  Male | 43 | 56 | 48 | 49 | 196

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1 Response [L] After 4 Weeks of Treatment
Description: Trough FEV1 (Forced expiratory volume in 1 second) was defined as the mean of the two FEV1 values (performed at 1 h and 10 min prior to study medication inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FEV1 response was defined as the change from baseline in trough FEV1. Baseline FEV1 was defined as the mean of the 2 pre-treatment FEV1 values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on ANCOVA with terms for baseline, treatment, and centre (centre random, all other effects fixed).
Time Frame: Baseline and 4 weeks
Population: Full Analysis Set (FAS). The FAS consisted of all patients who received at least 1 dose of study medication and had baseline data (pre-treatment at the end of the 2-week baseline) for at least 1 efficacy endpoint. For this trial all randomized and treated patients were included in the FAS.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L | 0.110 (0.021) | 0.134 (0.021) | 0.143 (0.020) | 0.168 (0.021)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.3791, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.029 to 0.076], Standard Error of Mean 0.027 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.2133, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.019 to 0.085], Standard Error of Mean 0.027 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p = 0.0337, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.057, 95% CI 2-sided [0.004 to 0.110], Standard Error of Mean 0.027 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

2. Secondary Outcome: Trough FEV1 Response [L] After 1 and 2 Weeks of Treatment.
Description: Trough FEV1 (forced expiratory volume in 1 second) was defined as the mean of the 2 FEV1 values (performed at 1 h and 10 min prior to study medication inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FEV1 response was defined as the change from baseline in trough FEV1. Baseline FEV1 was defined as the mean of the 2 pre-treatment FEV1 values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 15.
Time Frame: Baseline, 1 week and 2 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 8 | 0.093 (0.020) | 0.149 (0.020) | 0.154 (0.019) | 0.166 (0.020)
  Day 15 | 0.099 (0.020) | 0.141 (0.020) | 0.159 (0.020) | 0.154 (0.021)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.1163, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.010 to 0.093], Standard Error of Mean 0.026 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0224, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.060, 95% CI 2-sided [0.009 to 0.111], Standard Error of Mean 0.026 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p = 0.0380, ANCOVA — Type I error was controlled by a closed stepwise procedure; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.055, 95% CI 2-sided [0.003 to 0.107], Standard Error of Mean 0.026 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

3. Secondary Outcome: Trough FVC Response [L] After 1, 2 and 4 Weeks of Treatment
Description: Trough FVC (forced vital capacity) was defined as the mean of the 2 FVC values (performed at 1 h and 10 min prior to study medication inhalation) at the end of the dosing interval, 24 hours post-drug administration. Trough FVC response was defined as the change from baseline in trough FVC. Baseline FVC was defined as the mean of the 2 pre-treatment FVC values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: Baseline, 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 8 | 0.156 (0.033) | 0.215 (0.033) | 0.265 (0.032) | 0.275 (0.033)
  Day 15 | 0.171 (0.034) | 0.196 (0.034) | 0.280 (0.033) | 0.285 (0.034)
  Day 29 | 0.189 (0.036) | 0.191 (0.036) | 0.288 (0.036) | 0.306 (0.037)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.9573, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.002, 95% CI 2-sided [-0.089 to 0.094], Standard Error of Mean 0.047 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0321, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.099, 95% CI 2-sided [0.009 to 0.189], Standard Error of Mean 0.046 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p = 0.0125, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.117, 95% CI 2-sided [0.025 to 0.209], Standard Error of Mean 0.047 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

4. Secondary Outcome: FEV1 AUC(0-3h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment
Description: Response is defined as change from the baseline value. AUC(0-3h) (area under the curve) was calculated as the area under the curve from 0 to 3 hours on the various test days using the trapezoidal rule, divided by the full duration (3 hours) to report in litres. Baseline FEV1 was defined as the mean of the 2 pre-treatment FEV1 values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: 1 h and 10 min prior to inhalation and 5 min (only for week 1 and 2), 30 min, 1 h, 2 h and 3 h after inhalation at baseline and after 1, 2 and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 1 | 0.161 (0.016) | 0.201 (0.016) | 0.229 (0.016) | 0.225 (0.016)
  Day 8 | 0.204 (0.024) | 0.289 (0.024) | 0.302 (0.023) | 0.315 (0.024)
  Day 15 | 0.201 (0.024) | 0.288 (0.024) | 0.305 (0.024) | 0.309 (0.025)
  Day 29 | 0.191 (0.023) | 0.276 (0.023) | 0.270 (0.022) | 0.316 (0.023)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0052, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.085, 95% CI 2-sided [0.026 to 0.145], Standard Error of Mean 0.030 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0086, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.079, 95% CI 2-sided [0.020 to 0.138], Standard Error of Mean 0.030 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.125, 95% CI 2-sided [0.066 to 0.185], Standard Error of Mean 0.030 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

5. Secondary Outcome: FVC AUC(0-3h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment.
Description: FVC (forced vital capacity) AUC(0-3h) response is defined as change from the baseline value. AUC(0-3h) was calculated as the area under the curve from 0 to 3 hours on the various test days using the trapezoidal rule, divided by the full duration (3 hours) to report in litres. Baseline FVC was defined as the mean of the 2 pre-treatment FVC values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: as for outcome 4
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 1 | 0.268 (0.032) | 0.331 (0.032) | 0.413 (0.031) | 0.410 (0.032)
  Day 8 | 0.310 (0.042) | 0.441 (0.042) | 0.493 (0.041) | 0.537 (0.042)
  Day 15 | 0.327 (0.044) | 0.437 (0.044) | 0.513 (0.043) | 0.554 (0.044)
  Day 29 | 0.308 (0.043) | 0.424 (0.043) | 0.492 (0.043) | 0.547 (0.044)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0384, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.116, 95% CI 2-sided [0.006 to 0.225], Standard Error of Mean 0.056 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0009, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.184, 95% CI 2-sided [0.076 to 0.292], Standard Error of Mean 0.055 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.239, 95% CI 2-sided [0.130 to 0.349], Standard Error of Mean 0.056 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

6. Secondary Outcome: PEF AUC(0-3h) Response [L/Min] After First Administration and After 1, 2 and 4 Weeks of Treatment.
Description: PEF (peak expiratory flow rate L/min) AUC(0-3h) response is defined as change from the baseline value. AUC(0-3h) will be calculated as the area under the curve from 0 to 3 hours on the various test days using the trapezoidal rule, divided by the full duration (3 hours) to report in litres/min. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: as for outcome 4
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L/min
  Day 1 | 21.973 (3.596) | 35.738 (3.614) | 35.350 (3.533) | 40.027 (3.646)
  Day 8 | 29.701 (4.966) | 52.816 (4.973) | 49.722 (4.875) | 53.448 (5.025)
  Day 15 | 32.108 (5.115) | 54.527 (5.130) | 53.829 (5.022) | 54.289 (5.180)
  Day 29 | 29.734 (4.889) | 52.091 (4.912) | 48.503 (4.802) | 56.688 (4.956)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0010, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 22.357, 95% CI 2-sided [9.057 to 35.657], Standard Error of Mean 6.760 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0053, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 18.769, 95% CI 2-sided [5.613 to 31.924], Standard Error of Mean 6.687 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 26.954, 95% CI 2-sided [13.565 to 40.343], Standard Error of Mean 6.805 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

7. Secondary Outcome: FEV1 AUC(0-6h) Response [L] After 4 Weeks of Treatment
Description: FEV1 (forced expiratory volume in 1 second) AUC(0-6h) response is defined as change from the baseline value. AUC(0-6h) will be calculated as the area under the curve from 0 to 6 hours on test day 29 using the trapezoidal rule, divided by the full duration (6 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on ANCOVA with terms for baseline, treatment, and centre (centre random, all other effects fixed).
Time Frame: 1 h and 10 min prior to inhalation at baseline and after 4 weeks and 30 min, 1 h, 2 h, 3 h, 4 h, 5 h and 6h after inhalation at baseline and after 4 weeks (Day 29)
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L | 0.194 (0.023) | 0.282 (0.023) | 0.280 (0.023) | 0.322 (0.024)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0048, ANCOVA; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.027 to 0.149], Standard Error of Mean 0.031 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0056, ANCOVA; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.025 to 0.146], Standard Error of Mean 0.031 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, and centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.128, 95% CI 2-sided [0.066 to 0.189], Standard Error of Mean 0.031 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

8. Secondary Outcome: FVC AUC(0-6h) Response [L] After 4 Weeks of Treatment
Description: FVC (forced vital capacity) AUC(0-6h) response is defined as change from the baseline value. AUC(0-6h) will be calculated as the area under the curve from 0 to 6 hours on test day 29 using the trapezoidal rule, divided by the full duration (6 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: as for outcome 7
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L | 0.309 (0.044) | 0.429 (0.044) | 0.492 (0.043) | 0.547 (0.044)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0332, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.120, 95% CI 2-sided [0.010 to 0.230], Standard Error of Mean 0.056 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0011, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.183, 95% CI 2-sided [0.074 to 0.292], Standard Error of Mean 0.055 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.238, 95% CI 2-sided [0.128 to 0.349], Standard Error of Mean 0.056 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

9. Secondary Outcome: PEF AUC(0-6h) Response [L] After 4 Weeks of Treatment
Description: PEF (peak expiratory flow rate L/min) AUC(0-6h) response is defined as change from the baseline value. AUC(0-6h) will be calculated as the area under the curve from 0 to 6 hours on test day 29 using the trapezoidal rule, divided by the full duration (6 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: as for outcome 7
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L | 30.576 (4.933) | 53.443 (4.956) | 50.319 (4.845) | 58.368 (5.001)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0009, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 22.867, 95% CI 2-sided [9.462 to 36.272], Standard Error of Mean 6.813 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0036, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 19.743, 95% CI 2-sided [6.484 to 33.002], Standard Error of Mean 6.739 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 27.793, 95% CI 2-sided [14.298 to 41.287], Standard Error of Mean 6.859 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

10. Secondary Outcome: FEV1 Peak(0-3h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment
Description: FEV1 (forced expiratory volume in 1 second) peak(0-3h) is the maximum post-dose value during the first 3 hours after first administration and after 1, 2 and 4 weeks of treatment. Response is defined as change from the baseline value. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: 5 min (only for week 1 and 2), 30 min, 1 h, 2 h and 3 h after inhalation at baseline and after 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 1 | 0.249 (0.019) | 0.284 (0.019) | 0.311 (0.019) | 0.321 (0.019)
  Day 8 | 0.276 (0.025) | 0.359 (0.025) | 0.378 (0.024) | 0.397 (0.025)
  Day 15 | 0.276 (0.026) | 0.361 (0.026) | 0.391 (0.026) | 0.386 (0.027)
  Day 29 | 0.266 (0.024) | 0.353 (0.024) | 0.348 (0.024) | 0.410 (0.024)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0079, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.088, 95% CI 2-sided [0.023 to 0.152], Standard Error of Mean 0.033 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0120, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.082, 95% CI 2-sided [0.018 to 0.146], Standard Error of Mean 0.032 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.144, 95% CI 2-sided [0.080 to 0.209], Standard Error of Mean 0.033 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

11. Secondary Outcome: FVC Peak(0-3h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment
Description: FVC (forced vital capacity) peak(0-3h) is the maximum post-dose value during the first 3 hours after first administration and after 1, 2 and 4 weeks of treatment. Response is defined as change from the baseline value. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: as for outcome 10
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 1 | 0.428 (0.037) | 0.476 (0.037) | 0.576 (0.036) | 0.583 (0.037)
  Day 8 | 0.437 (0.043) | 0.560 (0.043) | 0.615 (0.042) | 0.690 (0.043)
  Day 15 | 0.465 (0.047) | 0.586 (0.047) | 0.648 (0.046) | 0.697 (0.047)
  Day 29 | 0.431 (0.045) | 0.562 (0.045) | 0.634 (0.044) | 0.696 (0.046)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0296, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.131, 95% CI 2-sided [0.013 to 0.249], Standard Error of Mean 0.060 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0007, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.204, 95% CI 2-sided [0.087 to 0.320], Standard Error of Mean 0.059 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.265, 95% CI 2-sided [0.147 to 0.383], Standard Error of Mean 0.060 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

12. Secondary Outcome: PEF Peak(0-3h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment
Description: PEF (peak expiratory flow rate L/min) peak(0-3h) is the maximum post-dose value during the first 3 hours after first administration and after 1, 2 and 4 weeks of treatment. Response is defined as change from the baseline value. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: as for outcome 10
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
L
  Day 1 | 43.051 (4.445) | 53.801 (4.474) | 53.853 (4.370) | 62.360 (4.510)
  Day 8 | 47.819 (5.213) | 69.792 (5.227) | 69.254 (5.118) | 73.828 (5.279)
  Day 15 | 48.129 (6.897) | 79.890 (6.930) | 71.916 (6.775) | 73.886 (6.992)
  Day 29 | 47.104 (5.088) | 70.519 (5.114) | 65.800 (4.999) | 76.461 (5.159)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0010, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 23.414, 95% CI 2-sided [9.529 to 37.300], Standard Error of Mean 7.057 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0078, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 18.695, 95% CI 2-sided [4.961 to 32.430], Standard Error of Mean 6.981 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p < 0.0001, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 29.357, 95% CI 2-sided [15.379 to 43.335], Standard Error of Mean 7.105 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

13. Secondary Outcome: FEV1 and PEF (Unsupervised) AUC(0-6h) Response [L] After First Administration and After 1, 2 and 4 Weeks of Treatment
Description: AUC(0-6h) for FEV1, and PEF (unsupervised) were not studied because the pertinent information from the unsupervised pulmonary function tests was for the time interval from 9 to 12 hours post-dosing.
Time Frame: After first administration, 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: FEV1 (Unsupervised) AUC(6-12h) Response [L] After First Administration and 1,2 and 4 Weeks of Treatment
Description: FEV1 (forced expiratory volume in 1 second) AUC(6-12h) response is defined as change from the baseline value. AUC(6-12h) will be calculated as the area under the curve from 6 to 12 hours on the various test days using the trapezoidal rule, divided by the full duration (6 hours) to report in litres. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on ANCOVA with terms for baseline, treatment, and centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: 6 h, 9 h and 12 h after inhalation at baseline and after 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 87 | 88 | 86 | 83
L
  Day 1 | 0.143 (0.031) | 0.181 (0.031) | 0.209 (0.031) | 0.175 (0.032)
  Day 8 | 0.169 (0.035) | 0.203 (0.035) | 0.219 (0.035) | 0.172 (0.036)
  Day 15 | 0.142 (0.038) | 0.197 (0.038) | 0.205 (0.038) | 0.169 (0.039)
  Day 29 | 0.145 (0.034) | 0.189 (0.034) | 0.193 (0.034) | 0.180 (0.035)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.3517, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.044, 95% CI 2-sided [-0.049 to 0.138], Standard Error of Mean 0.048 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.3171, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.046 to 0.143], Standard Error of Mean 0.048 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p = 0.4654, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 0.035, 95% CI 2-sided [-0.060 to 0.130], Standard Error of Mean 0.048 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

15. Secondary Outcome: PEF (Unsupervised) AUC(6-12h) Response [L/Min] After First Administration and 1,2 and 4 Weeks of Treatment
Description: PEF (peak expiratory flow rate L/min) AUC(6-12h) response is defined as change from the baseline value. AUC(6-12h) will be calculated as the area under the curve from 6 to 12 hours on the various test days using the trapezoidal rule, divided by the full duration (6 hours) to report in litres/min. Baseline was defined as the mean of the 2 pre-treatment values measured at Visit 2 (-1 h and -10 min) prior to administration of the first dose of study medication.
  The means are adjusted, based on ANCOVA with terms for baseline, treatment, and centre (centre random, all other effects fixed).
  Comparisons between groups are presented for Day 29.
Time Frame: 6 h, 9 h and 12 h after inhalation at baseline and after 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 87 | 88 | 86 | 83
L/min
  Day 1 | 29.261 (5.245) | 41.838 (5.197) | 45.179 (5.253) | 41.852 (5.360)
  Day 8 | 30.139 (5.690) | 47.625 (5.643) | 48.503 (5.704) | 47.924 (5.819)
  Day 15 | 27.512 (5.680) | 42.179 (5.627) | 52.249 (5.688) | 45.798 (5.803)
  Day 29 | 28.396 (5.469) | 41.502 (5.438) | 48.212 (5.497) | 47.289 (5.606)
Statistical Analysis 1: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/2 μg; Test type: Superiority or Other; p = 0.0899, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 13.106, 95% CI 2-sided [-2.055 to 28.267], Standard Error of Mean 7.704 — 2 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 2: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/5 μg; Test type: Superiority or Other; p = 0.0111, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 19.817, 95% CI 2-sided [4.549 to 35.084], Standard Error of Mean 7.759 — 5 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium
Statistical Analysis 3: Comparison: 5 µg Tiotropium vs Tiotropium+Olodaterol 5/10 μg; Test type: Superiority or Other; p = 0.0166, ANCOVA; terms for baseline, treatment, centre (centre random, all other effects fixed); Mean Difference (Final Values) = 18.893, 95% CI 2-sided [3.458 to 34.329], Standard Error of Mean 7.844 — 10 µg Olodaterol + 5 µg Tiotropium minus 5 µg Tiotropium

16. Secondary Outcome: Weekly Mean Pre-dose Morning PEF [L/Min]
Description: The patient will record twice daily peak flow measurements using an Asthma Monitor®Am2+ (AM2+) device. Morning measurements will be performed immediately upon arising after the patient has cleared out mucus, prior to administration of trial and/or rescue medication.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: Throughout the 4 week treatment period
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 89 | 88 | 90 | 83
L/min
  Week 1 | 227.81 (3.198) | 244.43 (3.208) | 248.84 (3.174) | 248.76 (3.310)
  Week 2 | 228.57 (3.401) | 240.87 (3.415) | 249.99 (3.377) | 247.77 (3.524)
  Week 3 | 228.82 (3.663) | 239.61 (3.684) | 249.39 (3.639) | 248.33 (3.800)
  Week 4 | 226.49 (3.678) | 234.14 (3.699) | 249.17 (3.654) | 247.30 (3.816)

17. Secondary Outcome: Weekly Mean Evening PEF [L/Min]
Description: The patient will record twice daily peak flow measurements using an AM2+ device. The evening measurement will be performed at bedtime.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: Throughout the 4 weeks treatment period
Population: Full Analysis Set.
Measure: Mean (Standard Error); unit: L/min
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 89 | 88 | 92 | 84
L/min
  Week 1 | 249.10 (3.419) | 260.86 (3.425) | 267.47 (3.360) | 268.58 (3.510)
  Week 2 | 247.10 (3.804) | 260.73 (3.814) | 267.31 (3.738) | 266.40 (3.909)
  Week 3 | 249.78 (3.765) | 258.20 (3.791) | 268.16 (3.702) | 265.67 (3.884)
  Week 4 | 246.77 (3.777) | 253.12 (3.803) | 266.61 (3.714) | 265.50 (3.896)

18. Secondary Outcome: Weekly Mean Number of Occasions of Rescue Therapy Used Per Day
Description: The means are adjusted, Based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: Throughout the 4 weeks treatment period
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: occasion(s)
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 89 | 89 | 92 | 84
occasion(s)
  Week 1 | 1.905 (0.155) | 1.512 (0.155) | 1.504 (0.152) | 1.669 (0.159)
  Week 2 | 1.784 (0.178) | 1.610 (0.177) | 1.476 (0.175) | 1.477 (0.182)
  Week 3 | 1.947 (0.183) | 1.650 (0.182) | 1.492 (0.180) | 1.563 (0.187)
  Week 4 | 2.017 (0.172) | 1.615 (0.172) | 1.602 (0.169) | 1.482 (0.176)

19. Secondary Outcome: Physician's Global Evaluation
Description: Measured a 8-point scale, from 1 (poor) to 8 (excellent), as judged by the physician, over 4 weeks of treatment.
  The physician made a global evaluation at the end of the Baseline Period (Test Day 1) and at each visit thereafter. These assessments were made prior to pulmonary function testing and reflected the physician's opinion of the patient's overall clinical condition. This evaluation was based on the need for concomitant medication, number and severity of COPD exacerbations since the last visit, severity of cough, ability to exercise, amount of wheezing, and other relevant clinical observations.
  The means are adjusted, based on an ANCOVA with terms for baseline, treatment, centre (centre random, all other effects fixed).
Time Frame: 1 week, 2 weeks and 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 92 | 88
units on a scale
  Day 8 | 5.139 (0.102) | 5.102 (0.102) | 5.185 (0.100) | 5.149 (0.102)
  Day 15 | 5.272 (0.113) | 5.130 (0.113) | 5.382 (0.111) | 5.104 (0.113)
  Day 29 | 5.264 (0.115) | 5.295 (0.115) | 5.447 (0.113) | 5.252 (0.115)

20. Secondary Outcome: Patient's Global Rating
Description: Patient's Global Rating at the end of the 4 week treatment period.
  Patients rated their health (respiratory condition) at Day 29 (compared to the day before they commenced treatment with study medication) on a 7-point scale as "very much better (1), much better (2), a little better (3), no change (4), a little worse (5), much worse (6), or very much worse (7)". The assessment was made prior to pulmonary function testing and all other study procedures. The Patient's Global Rating was also completed before the Physician's Global Evaluation.
  The means are adjusted, based on an ANCOVA with terms for treatment, centre (centre random, treatment effect fixed).
Time Frame: 4 weeks
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: units on a patient's global rating score
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 86 | 87 | 90 | 84
units on a patient's global rating score | 2.866 (0.112) | 2.598 (0.111) | 2.368 (0.109) | 2.377 (0.113)

21. Secondary Outcome: Clinically Significant Anormalities (Laboratory Data); Marked Changes From Baseline for Vital Signs, Notable Change in ECG and New Onset of ECG Abnormalities
Description: Possible clinically significant anormalities (laboratory data); marked changes from baseline for vital signs, notable change in ECG and new onset of ECG abnormalities. New abnormal findings or worsening of baseline conditions were reported as Adverse Events (AEs).
  All AEs with an onset after the first dose of study medication up to 21 days after the last dose of study medication were to have been assigned to the Treatment Period.
Time Frame: From first dose up to 21 days after last dose of study medication.
Population: Treated Set.
Measure: Number; unit: participants
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 90 | 89 | 93 | 88
participants | 1 | 0 | 0 | 0

22. Secondary Outcome: Cmax,ss Olodaterol [pg/mL]
Description: Maximum measured concentration of Olodaterol in plasma at steady state (Cmax,ss) after 4 weeks of treatment.
  No results displayed for Tiotropium+Olodaterol 5/2 μg because there were zero total participants analyzed for this outcome measure.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of PK or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 42 | 59
pg/mL | 4.39 (49.2) | 6.87 (56.1)

23. Secondary Outcome: Tmax,ss Olodaterol [h]
Description: Time from last dosing to maximum concentration of Olodaterol in plasma at steady state (tmax,ss) after 4 weeks treatment.
  No results displayed for Tiotropium+Olodaterol 5/2 μg because there were zero total participants analyzed for this outcome measure.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients.
Measure: Median (Full Range); unit: hours
Arm/Group | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 42 | 59
hours | 0.167 [0.083 to 0.917] | 0.183 [0.067 to 1.070]

24. Secondary Outcome: AUC(0-1h,ss) Olodaterol [pg*h/mL]
Description: Area under the concentration-time curve of Olodaterol in plasma at steady state (AUC(0-1h,ss)) from 0 to 1 hour post dosing after 4 weeks of treatment.
  No results displayed for Tiotropium+Olodaterol 5/2 μg because there were zero total participants analyzed for this outcome measure.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 28 | 52
pg*h/mL | 3.97 (49.4) | 5.82 (50.5)

25. Secondary Outcome: Cmax,ss Tiotropium [pg/mL]
Description: Maximum measured concentration of Tiotropium in plasma at steady state (Cmax,ss) after 4 weeks treatment.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 78 | 78 | 73 | 73
pg/mL | 13.3 (75.3) | 13.9 (64.7) | 12.4 (69.7) | 14.4 (69.1)

26. Secondary Outcome: Tmax,ss Tiotropium [h]
Description: Time from last dosing to maximum concentration of Tiotropium in plasma at steady state (tmax,ss) after 4 weeks of treatment.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients.
Measure: Median (Full Range); unit: hours
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 73 | 78 | 78 | 73
hours | 0.133 [0.050 to 1.000] | 0.100 [0.017 to 0.983] | 0.083 [0.067 to 0.917] | 0.133 [0.050 to 1.000]

27. Secondary Outcome: AUC(0-3h,ss) Tiotropium [pg*h/mL]
Description: Area under the concentration-time curve of Tiotropium at steady state (AUC(0-3h,ss)) from 0 to 3 hours post dosing after 4 weeks of treatment.
Time Frame: Pre-dose, 5 min, 10 min, 20 min, 40 min, 1 h, 3 h, and 6 h after the last dose.
Population: Evaluable patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Number analyzed (Participants) | 58 | 59 | 56 | 50
pg*h/mL | 21.8 (42.8) | 21.9 (45.3) | 21.9 (47.9) | 21.0 (42.9)

ADVERSE EVENTS:
Time Frame: From first dose up to 21 days after last dose of study medication, upto 86 days.
Description: At each visit, all AEs, regardless of causality, were recorded on the AE e-CRF page after review of the e-Diary and discussion with the patient. Adverse events were recorded on the eCRFs as non-serious or SAEs.
Arm/Group | 5 µg Tiotropium | Tiotropium+Olodaterol 5/2 μg | Tiotropium+Olodaterol 5/5 μg | Tiotropium+Olodaterol 5/10 μg
Serious Adverse Events (participants affected / at risk) | 2/90 | 3/89 | 1/93 | 0/88
Other Adverse Events (participants affected / at risk) | 0/90 | 0/89 | 0/93 | 0/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 5 µg Tiotropium (N=90) | Tiotropium+Olodaterol 5/2 μg (N=89) | Tiotropium+Olodaterol 5/5 μg (N=93) | Tiotropium+Olodaterol 5/10 μg (N=88)
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.